CLINICAL TRIAL: NCT01725516
Title: Effect of Myofascial Release Technique on Reducing Symptoms in Patients With Chronic Disc Protrusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Other Study IDs: 90-01-06-4234
Record Dates: First submitted 2012-11-13; First posted 2012-11-14 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2011-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Myofascial release technique (Experimental)
  Interventions: Procedure: Myofascial release technique

INTERVENTIONS:
Procedure: Myofascial release technique

SUMMARY:
The purpose of this study is to determine whether myofascial release technique are effective in the treatment of low back pain due to lumbar disc herniation.

ELIGIBILITY:
Inclusion Criteria:

* lumbar disc herniation
* Muscular trriger points
* independent ambulated patients

Exclusion Criteria:

* Neoplasm
* Lumbar surgery history
* fracture
* inflammatory disease

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult

PRIMARY OUTCOMES:
Pain

SECONDARY OUTCOMES:
Oswestry Disability Index